CLINICAL TRIAL: NCT03881293
Title: Effects of Topical Lidocaine During Urodynamic Testing In Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristine Zinkgraf (Other)
Collaborators: Medical College of Wisconsin (Other); WomenConnected (Unknown)
Responsible Party: Sponsor-Investigator, Kristine Zinkgraf, Advanced Practice Nurse, ProHealth Care, Inc
Organization: ProHealth Care, Inc (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IRB#12-09
Record Dates: First submitted 2019-02-15; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Urinary Stress Incontinence; Pain
Keywords: urodynamics; women; lidocaine gel
MeSH Terms: conditions — Urinary Incontinence, Stress; Pain | interventions — Lidocaine; Gels

STUDY DESIGN:
Intervention Model Description: Double Blinded Randomized Control Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Lubricant Gel (Placebo Comparator): 5 ml water-soluble gel instilled transurethrally ten minutes prior to catheter insertion
  Interventions: Drug: water soluble lubricant
- Lidocaine 2% Gel (Active Comparator): 5 ml lidocaine 2% gel instilled transurethrally ten minutes prior to catheter insertion
  Interventions: Drug: lidocaine 2% gel

INTERVENTIONS:
Drug: lidocaine 2% gel — Transurethral instillation of 5 ml lidocaine 2% gel
  Arms: Lidocaine 2% Gel
Drug: water soluble lubricant — Transurethral instillation of 5 ml water soluble lubricant
  Arms: Placebo Lubricant Gel

SUMMARY:
Urodynamic testing is used to help diagnose causes of urinary incontinence and voiding dysfunction. The purpose of the urodynamic test is to gain insight into the patient's urinary symptoms and assist in making a diagnosis. Catheter insertion and manipulation during the test can be uncomfortable for the patient. Lidocaine gel has not been used routinely during urodynamic testing. However, it is used routinely during outpatient cystoscopy and with any urethral catheterization. The investigators proposed that lidocaine numbing gel could be used without compromising test findings.

The study included 110 adult women. The purpose was:

1. Determine whether the use of topical lidocaine during urodynamic testing decreases patient discomfort during the procedure.
2. Evaluate whether the use of topical lidocaine affects the urodynamic results.

DETAILED DESCRIPTION:
Topical Lidocaine For Urodynamic Testing: A Double Blinded Randomized Control Trial

Hypothesis / aims of study

1. Determine whether the use of topical lidocaine during urodynamic testing decreases patient discomfort during the procedure.
2. Evaluate whether the use of topical lidocaine affects the urodynamic results.

Study design, materials and methods The hospital IRB approved the study. Women with symptoms of stress urinary incontinence (SUI) scheduled for a urodynamic study (UDS) were eligible to participate. Women presenting with predominant overactive bladder symptoms were excluded. Participants were randomized on the day of the procedure using Random Allocation Software Version 1.0. All were blinded to the study arms until completion of final data analysis. Participant randomization assignment was known only to an independent research nurse and the dispensing pharmacist. The study consisted of transurethral administration of 5 ml lidocaine 2% gel or surgilube gel, in the study and control arms, respectively, 10 minutes before catheter insertion. Prior to testing, a 24 hour bladder diary and the Pelvic Floor Distress Inventory - Short Form 20 were completed. During the UDS participants were asked for sensory information including desire to void and maximal cystometric capacity (MCC). Urethral pressure profiles were obtained at an infused volume of 200 ml. Provocative measures were performed to assess SUI. Using a Likert scale, pain was assessed prior to and after catheter insertion, after performing the urethral pressure profile, and at the completion of the study. The primary outcome; pain after urethral pressure profile (UPP), was compared between the two groups. Comparisons of the bladder diary and UDS results were made between study and control arms individually and in-between groups.

Statistical methods The effect of lidocaine on patient pain as reported during multiple time-points during the UDS was evaluated using repeated measures analysis via mixed effects regression with a random patient-specific intercept. This approach allows the evaluation of the overall pain experience, as well as baseline-adjusted comparison at individual time-points. Comparisons were done using t-tests for continuous variables, Chi-squared test for categorical variables, Wilcoxon rank-sum test, Lin's Concordance Correlation Coefficient (CCC), and a z-test. The CCC provides a generalization of Pearson's correlation coefficient that measures how well the data align with the diagonal representing equal values for the two measurements (as opposed to any straight line). Agreement is stronger than correlation. Specifically, the agreement between mean void volume and volume at strong desire, as well as between maximum void volume and volume at MCC were computed separately for each study group. The CCC values were compared between the study groups using a z-test. Power calculations determined a total sample size of 110 participants was needed to detect significant differences between the groups with at least 94% statistical power.

ELIGIBILITY:
Inclusion Criteria:

Women with complaint of stress urinary incontinence who were scheduled for a urodynamic test Patients with symptomatic pelvic organ prolapse if they also had stress incontinence symptoms.

Community dwelling elderly patients who were able to provide their own history and were able to sign for themselves

Exclusion Criteria:

Patients who were unable to provide their own consent Patients who are allergic to lidocaine Children and pregnant patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 110 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in pain immediately after urethral pressure profilometry | Pain was assessed immediately after urethral pressure profilometry was performed
  Patient rated pain using Likert Scale of 0-10 (0 is no pain and 10 is worst pain)

SECONDARY OUTCOMES:
Demonstration of stress urinary incontinence during the urodynamic test | During the urodynamic test
  Ability to demonstrate stress urinary incontinence during the urodynamic test
Perception of bladder filling | During the urodynamic test
  Correlation of maximal cystometric capacity on urodynamic test and maximal voided volume on bladder diary

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Stevenson, MD, Principal Investigator — ProHealth Care

IPD SHARING:
Plan to Share IPD: No